CLINICAL TRIAL: NCT05917392
Title: Effects of Polyphenol and Lactobacillus Rhamnosus Supplementation in Fermented Vegetables (Kimchi) on Gut Microbiota, DNA Methylation and Serum Proteomes in Overweight and Obese Women
Brief Title: Effects of Kimchi Supplementation on Gut Microbiota, DNA Methylation and Serum Proteomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: COA. MURA2023/127
Record Dates: First submitted 2023-05-21; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Obesity
Keywords: DNA methylation; proteomic; microbiota
MeSH Terms: conditions — Obesity | interventions — Dietary Supplements; Probiotics; Polyphenols

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supplementation-standard (Active Comparator): Supplementation with Kimchi 50 gram daily for two months
  Interventions: Dietary Supplement: Fermented Vegetables (Kimchi) supplementation
- Supplementation with probiotic (Experimental): Supplementation with Kimchi plus LGG 50 gram daily for two months
  Interventions: Dietary Supplement: probiotic
- Supplementation with polyphenol (Experimental): Supplementation with Kimchi plus polyphenol 50 gram daily for two months
  Interventions: Dietary Supplement: polyphenol

INTERVENTIONS:
Dietary Supplement: Fermented Vegetables (Kimchi) supplementation — Fermented Vegetables (Kimchi) supplementation with 50 gm daily for two months and effects of DNA methylation, serum proteome and microbiota
  Other Names: Kimchi supplementation
  Arms: Supplementation-standard
Dietary Supplement: probiotic — Supplementation with Kimchi plus LGG 50 grams daily for two months
  Arms: Supplementation with probiotic
Dietary Supplement: polyphenol — Supplementation with Kimchi plus polyphenol 50 grams daily for two months
  Arms: Supplementation with polyphenol

SUMMARY:
Participants will ask to answer questionnaire related to general characteristic, lifestyle, dietary pattern and undergo physical examination and measurement of body composition. The subjects will be divided into 2 groups: healthy control and intervention. The intervention group was divided into 3 subgroups: the fermented vegetable (kimchi) group, the kimchi supplemented with polyphenol (Vitexin) group, or the kimchi supplemented with probiotic (Lactobacillus rhamnosus) group. The intervention group will be instructed to consume 1 pack of kimchi per day (50 g/pack) with lunch for 2 months.

DETAILED DESCRIPTION:
The subjects will be divided into 2 groups: healthy control and intervention. The intervention group was divided into 3 subgroups: the fermented vegetable (kimchi) group, the kimchi supplemented with polyphenol (Vitexin) group, or the kimchi supplemented with probiotic (Lactobacillus rhamnosus) group. The intervention group will be instructed to consume 1 pack of kimchi per day (50 g/pack) with lunch for 2 months. During the study, participants will be strongly encouraged to avoid consuming prebiotics or probiotic supplements, as well as foods such as yogurt, sour milk, fermented vegetables, and fermented fruits, especially 2 weeks before the blood and fecal examination. Compliance will be assessed by monitoring product side effects through follow-up phone calls every week to check on participants' symptoms and assessing the number of sachets or packs they actually consume.

ELIGIBILITY:
Inclusion Criteria: for the intervention group

* age 35-50 years, BMI of ≥23 kg/m2, presence or absence of metabolic syndrome (not treated by medication) according to the National Cholesterol Education Program (NCEP ATPIII 2007), in collaboration with the International Diabetes Federation (IDF) and the World Health Organization (WHO), metabolic syndrome

Exclusion Criteria:for the intervention group

* participants declined or withdrew, history of taking antibiotics in the 12 weeks prior to the project, history of using prebiotics or probiotic supplements on a regular basis, history of eating foods in these groups regularly, including yogurt, sour milk, fermented vegetables, and fermented fruits, history of taking drugs or weight loss products in the previous 6 months, history of diarrhea or constipation regularly, history of cure for ulcerative colitis, history of underlying disease that requires continuous medication, history of taking laxatives regularly, history of severe gastrointestinal disease, and history of illnesses such as thyroid disease, cancer, autoimmune diseases, kidney disease and hypertension etc.

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
ฺBMI | 2 months
  changes in BMI for evaluating obesity at 2 months from baseline
gut bacterial flora | 2 months
  Changes and differences of the gut bacterial flora will be addressed in detail, e.g. changes in concentration of specific bacterial groups (e.g. Lactobacillus) before and after the intervention period.

SECONDARY OUTCOMES:
DNA methylation of inflammation and anti-inflammation gene | 2 months
  changes in methylation (hypomethylation and hypermethylation)
Serum proteome | 2 months
  changes in protein expression (up and dow-regulation)

OTHER OUTCOMES:
The differences between the treatment groups and the non-obese group for exploratory variables | baseline
  Changes in blood biochemistry (lipid profile, inflammatory cytokine level), protein expression (up and dow-regulation), %methylation (hypomethylation and hypermethylation) and concentration of specific bacterial groups

CONTACTS AND LOCATIONS:
Overall Officials: Jintana Sirivarasai, Ph.D, Principal Investigator — Ramathibodi Hospital
Locations (1):
- Jintana Sirivarasai, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: starting 12 months after publication
Access Criteria: After summary data are published and others can access via journal website